CLINICAL TRIAL: NCT00472264
Title: An Exploratory Study To Investigate The Reproducibility Of Lung 18Fluoro-Deoxyglucose Positron Emission Tomography In Patients With Chronic Obstructive Airways Disease (COPD) In The Absence Of Anti-Inflammatory Treatments
Brief Title: A Study To Investigate The Ability To Use 18FDG PET Scanning To Monitor The Effectiveness Of New Drugs In COPD Patients
Status: Terminated | Type: Observational
Why Stopped: Study terminated on Nov 7, 2008 as a result of poor recruitment and changes in business priorities. The decision was not based on safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A9011012
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: methodology study, PET Imaging, COPD patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm study (Healthy volunteers & COPD subjects): A single arm study PET imaging is carried out twice during the first week of the study and again 4 weeks later in both Healthy volunteers and COPD subjects.
  Interventions: Procedure: PET imaging

INTERVENTIONS:
Procedure: PET imaging — Medical imaging assessment

SUMMARY:
It is hypothesised that there is a difference between the uptake of a radioactive substance ([18F]fluorodeoxyglucose (FDG)) in the lungs of patients with Chronic Obstructive Pulmonary Disease (COPD) and healthy volunteers.

DETAILED DESCRIPTION:
Single site, eligible subjects enrolled in order of presentation.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients:
* Subjects with a Body Mass Index (BMI) between 18-32 kg/m2.
* Patients with a diagnosis, for at least 6 months, of moderate to severe (Stage II - III) COPD as defined by the NIH/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2005 revision), whose disease has been stable for 3 months, and have not had a respiratory tract infection for 6 weeks prior to screening.
* Ability to be maintained off inhaled corticosteroids and other anti-inflammatory medications (e.g., theophylline) as required by the protocol
* Healthy Volunteers:
* Healthy volunteers should be age (+/- 5 years) and gender matched to the COPD subjects
* No history of asthma, COPD or other lung disease (including, sarcoidosis, pneumoconiosis, tuberculosis, lung surgery or resection, lung cancer, bronchitis).
* Free from clinically significant disease.

Exclusion Criteria:

* Exacerbation or hospitalisation for COPD within 3 months of screening, or more than twice during the preceding year.
* Use of oral corticosteroids in the 6 weeks prior to screen. (Patients who have been taking inhaled corticosteroids as maintenance COPD therapy are eligible provided the dose has remained stable for the previous 6 weeks and it is considered that they could tolerate withdrawal of inhaled corticosteroid for the duration of the study).
* A clearly documented history of adult asthma or other chronic respiratory disorders apart from COPD (e.g. clinically significant bronchiectasis, pulmonary fibrosis, pneumoconiosis).
* Previous history of bronchial carcinoma, or previous history of lung surgery (including lung resection, pleurodesis, open lung biopsy, video-assisted lung biopsy) or invasive lung procedure (e.g., bronchoscopy (with or without biopsy), bronchoalveolar lavage).
* Patients with a history of prior radiation exposure within the past year such that participation this study would put them over 5 rem for annual radiation exposure for research subjects.
* History or evidence, based upon a complete medical history, full physical examination, chest X-ray or clinical laboratory test results, of any other significant concomitant clinical disease that, in the opinion of the investigator, could interfere with the subject's safety or the conduct of this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 Moderate to Severe COPD patients and 8 age- and gender-matched Healthy Volunteer Subjects.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Uptake of FDG (Ki) at <1 and 4 weeks | <1 and 4 weeks

SECONDARY OUTCOMES:
BODE Index (Screening) | Screening
Chronic Respiratory Questionnaire (1week and 4 weeks) | <1 week and 4 weeks
Emphysema index (chest CT emphysema score) (Screening) | Screening
Airway wall area (as % total airway cross-sectional area) (chest CT assessment, see Appendix 3 for details) (1 week and 4 weeks) | <1 week and 4 weeks
Clinical COPD Questionnaire (Screening 1 week and 4 weeks) | Screening <1 week and 4 weeks
COPD GOLD Stage (screening) | Screening
Lung function indices (FEV1, FVC, FEV1/FVC, DLco) and lung volumes (TLC, IC, RV) (Screening 1 week and 4 weeks) | screening, <1 week and 4 weeks
St. George's Respiratory Questionnaire (screening) | Screening
Smoking history (screening) | Screening

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, St Louis, Missouri, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011012&StudyName=A%20Study%20To%20Investigate%20The%20Ability%20To%20Use%2018FDG%20PET%20Scanning%20To%20Monitor%20The%20Effectiveness%20Of%20New%20Drugs%20In%20COPD%20Patients